CLINICAL TRIAL: NCT04559243
Title: A Prospective, Multicenter Clinical Study of Percutaneous Left Atrial Appendage Closure as Secondary Prevention of Atrial Fibrillation-related Embolic Events in Patients With Atrial Fibrillation
Brief Title: Left Atrial Appendage Closure as Secondary Prevention of Atrial Fibrillation-related Embolic Events
Status: Recruiting | Type: Observational
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAAC-01
Record Dates: First submitted 2020-09-14; First posted 2020-09-22 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Non-valvular Atrial Fibrillation; Embolic Stroke
Keywords: AF-related embolic events; non-valvular atrial fibrillation; Left Atrial Appendage Closure
MeSH Terms: conditions — Embolic Stroke | interventions — Echocardiography; Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — After the surgey, the tests data will be collected during 8 visits when the subjects go back to the hospital.
  Other Names: Transesophageal Echocardiography

SUMMARY:
This clinical study is a prospective, multi-center, non-interventional study designed to investigate the safety and effectiveness of percutaneous LAA appendage closure by using LAmbre™ Left Atrial Appendage Occluder System. 579 patients with valvular AF complicated with previous AF-related embolic events (including ischemic stroke, TIA and systemic embolism) were enrolled at about 20 study sites nationwide. The baseline data, operation process and relevant follow-up information of subjects were recorded at 7 months after operation or before discharge and at 1, 3, 6, 12 and 24 months after operation.

DETAILED DESCRIPTION:
Study Population Patients with non-valvular atrial fibrillation and previous AF-related embolic events Purpose To assess the feasibility and safety of percutaneous LAA closure as secondary prevention for patients with non-valvular atrial fibrillation (NVAF) and previous atrial fibrillation (AF) related embolic events (including ischemic stroke, transient ischemic attack (TIA), and systemic embolism).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female;
* Patients who are able to understand the purpose of the study, voluntarily participate in and sign the informed consent form (ICF), and are willing to complete the follow-up as required by the protocol;
* Indications for left atrial appendage closure;
* Patients with non-valvular AF complicated with previous AF related embolic event and meeting one of the following conditions;

  1. HAS-BLED bleeding risk score ≥ 3 points;
  2. Not suitable for long-term oral anticoagulant therapy;
  3. Poor compliance with oral anticoagulants;
  4. CHA2DS2-VASc score ≧ 2 points;

Exclusion Criteria:

* Valvular AF (after moderate to severe mitral stenosis or mechanical valve replacement)
* Initial AF, reversible AF with clear cause
* Presence of adherent thrombus in the left atrium or left ventricular aneurysm thrombus
* ST elevation myocardial infarction, ≤ 3 months
* Grade-IV of Cardiac Function (NYHA)
* Allergy or contraindication to metal nitinol, aspirin, clopidogrel, heparin, and other anticoagulants
* Pregnant or with plan of pregnancy during the study
* Participation in another drug or medical device clinical trial or study that has not been completed
* Experience new stroke or TI within 30 days or major bleeding events within 14 days
* Contraindication to LAA closure or deemed unsuitable for study participation by the investigator
* Had a definite thromboembolic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation and previous AF-related embolic events
Sampling Method: Non-Probability Sample
Enrollment: 579 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of new ischemic stroke, systemic embolism, and cardiac death 12 months after operation | 12 months
  Ischemic stroke, systemic embolism, and cardiac death events
Incidence of major bleeding events (intracranial or gastrointestinal, or any bleeding requiring transfusion of ≥ 2 units of red blood cells) at 12 months after operation | 12 months
  Bleeding events

SECONDARY OUTCOMES:
Surgical success rate | 24 months
  Surgical success
Success rate of LAA closure at 3 months after operation | 3 months
  Successful LAA closure was defined as a residual shunt ≤ 3 mm by TEE or ICE after implantation of the LAA occluder.
The composite endpoint of new ischemic stroke, systemic embolism and cardiac death at 7 months after operation or before discharge and at 1, 3, 6 and 24 months after operation | 24 months
  Ischemic stroke, systemic embolism, and cardiac death events
(4)Perioperative (7 days after operation or before discharge) surgery-related complications | 7 days
  7 days after operation or pre-discharge procedure-related complications include but are not limited to stroke (ischemic and hemorrhagic stroke), systemic embolism, allergic reaction, gas embolism, pericardial effusion/cardiac tamponade requiring intervention, occluder detachment, occluder thrombosis (DRT), minor bleeding events (including but not limited to puncture site hematoma, non-major bleeding events), infection, arrhythmia, damage to blood vessels or organs on the implantation path and adjacent organs
Procedure-related complications during follow-up | 24 months
  Follow-up at 1, 3, 6, 12 and 24 months after operation for procedure-related complications, including all-cause death, stroke (ischemic and hemorrhagic stroke), cardiac perforation, pericardial effusion/cardiac tamponade requiring intervention, major bleeding events (intracranial or gastrointestinal, or any bleeding requiring transfusion of ≥ 2 units of red blood cells), occluder thrombosis (DRT), infection, systemic embolism, allergic reaction, arrhythmia, and other serious cardiovascular events requiring intervention or surgical treatment
Occluder defects during operation and in the 3rd month after operation | 3 months
  Including but not limited: Occluder displacement, Occluder detachment, Occluder breakage, Occluder damage, etc
Incidence rate of severe adverse events within 24 months after operation | 24 months
  including but not limited to all-cause death, events requiring hospitalization or prolongation of hospitalization, severe endocarditis requiring surgery, pericarditis, cardiac perforation, valvular injury, vascular or gas embolism events, occluder detachment/displacement, occluder fracture, occluder thrombosis (DRT), stroke events

CONTACTS AND LOCATIONS:
Overall Officials: Chenyang Jiang, Doctor, Principal Investigator — Sir Run Run Shaw Hospital; Jinhua Zhang, Doctor, Principal Investigator — Sir Run Run Shaw Hospital
Locations (5):
- China (5):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Songjiang District Central Hospital, Shanghai, Shanghai Municipality
  - Sichuan Mianyang 404 Hospital, Mianyang, Sichuan
  - The first Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided